CLINICAL TRIAL: NCT05380791
Title: Effect of Esophageal Contractile Reserve on Changes in Esophageal Motility and Symptoms After Anti-reflux Surgery in Patients With Gastroesophageal Reflux Disease
Brief Title: Effect of Esophageal Contractile Reserve on Changes in Esophageal Motility and Symptoms After ARS in Patients With GERD
Status: Recruiting | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice-President, Shandong University
Other Study IDs: 2022-SDU-QILU-008
Record Dates: First submitted 2022-04-21; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Esophageal Motility Disorders
Keywords: contraction reserve
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IEM in patients with GERD with normal MRS contraction: Esophageal motility determined by high resolution esophageal manometry and multiple rapid swallow (MRS) tests
  Interventions: Other: Follow-up visits
- IEM in patients with GERD with abnormal MRS contraction: Esophageal motility determined by high resolution esophageal manometry and multiple rapid swallow (MRS) tests
  Interventions: Other: Follow-up visits

INTERVENTIONS:
Other: Follow-up visits — Regular follow-up visits to record information about the patient's surgery and routine post-operative examinations
  Other Names: Questionnaire to assess symptoms and quality of life etc.

SUMMARY:
rapid swallow (MRS) can assess the contractile reserve capacity of the oesophageal body and identify and diagnose oesophageal motility disorders, but the impact of preoperative oesophageal reserve capacity on postoperative symptoms and motility in patients with GERD remains unclear. The aim of this study was to assess the effect of pre-operative oesophageal reserve capacity on post-reflux symptoms and motility in patients with GERD by using a high-resolution oesophageal manometry-based provocation test, MRS, to track pre-operative ineffective oesophageal motility (IEM).

DETAILED DESCRIPTION:
Lower oesophageal sphincter relaxation is an important cause of GERD and ineffective oesophageal motility may be associated with GERD, but the mechanism of oesophageal corporal motility disorders is unclear. High-resolution manometry (HRM) has shown to be more accurate than conventional manometry in assessing oesophageal motility, and can provide guidance for GERD surgery. The aim was to conduct a cohort study to investigate the yu'h of patients with preoperative esophageal motility disorders with or without esophageal reserve, based on the assessment of esophageal motility by high-resolution esophageal manometry to follow up changes in esophageal motility and symptoms in patients after anti-reflux surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Patients to be treated surgically for gastroesophageal reflux disease
* Ineffective esophageal motility diagnosed by high resolution esophageal manometry according to Chicago Classification version 4.0
* Obtaining Informed Consent

Exclusion Criteria:

* Previous other upper gastrointestinal surgery
* Pregnant women and other people with contraindications to surgery and tests
* Other specifically defined esophageal motility disorders, such as nutcracker esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to be treated surgically for gastroesophageal reflux disease. Ineffective esophageal motility diagnosed by high resolution esophageal according to Chicago Classification version 4.0(defined as ≥ 70% of swallows with weak contraction (distal contraction interval (DCI) between 100mmHg/s/cm and less than 450 mmHg/s/cm) or ≥ 50% of swallows with failed peristalsis Performance.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Effect of changes in oesophageal motility after anti-reflux surgery compared to pre-surgery | 2 year follow-up after anti-reflux surgery
  Using high resolution manometry to assess changes in oesophageal motility after anti-reflux surgery, compared to pre-surgery.

SECONDARY OUTCOMES:
Effect of changes of post-anti-reflux surgery symptoms | 2 year follow-up after anti-reflux surgery
  Reflux Symptom Questionnaire Assessment to assess the changes of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, phD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided